CLINICAL TRIAL: NCT01447563
Title: Bioavailability of Two Oral Formulations of Clopidogrel: A Randomized, Open Label, Single Dose, Two-Period, Crossover Comparison in Healthy Mexican Volunteers
Brief Title: Comparative Bioavailability Study of Two Oral Formulations of Clopidogrel
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Lourdes Garza Ocañas, Principal Investigator, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CLOPI Tabs No. 60-06
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Comparative Bioavailability of Clopidogrel Tablets
Keywords: Bioequivalence; Bioavailability
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel tablets 75mg (Experimental): subjects received a single 75 mg tablet of the reference formulation, given with 250 mL water
  Interventions: Drug: Clopidogrel bisulfate
- Clopidogrel (Experimental): subjects received a single 75 mg tablet of the test formulation, given with 250 mL water
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel bisulfate — subjects received a single 75 mg tablet of the reference formulation, given with 250 mL water
  Other Names: Plavix
  Arms: Clopidogrel tablets 75mg
Drug: Clopidogrel — subjects received a single 75 mg tablet of the test formulation, given with 250 mL water
  Arms: Clopidogrel

SUMMARY:
Background: Clopidogrel, a potent inhibitor of adenosine diphosphate-induced platelet activation, is widely used to prevent and reduce the risk of thrombotic events. Objective: the aim of the present study is to evaluate the bioequivalence of two oral formulations of 75 mg clopidogrel tablets. Method: The study is an open, randomized, single-dose, two-period crossover trial conducted on 32 healthy Mexican volunteers in a fasted state. A single oral dose of the test or reference drug will be followed by a 7 day washout period, after which subjects will receive the alternative formulation. Blood samples were collected up to 24 h after dosing. In order to determine bioequivalence, the plasma concentrations of clopidogrel carboxylic acid metabolite was determined using high-performance liquid chromatography-tandem mass spectrometry area under the plasma concentration time curve from zero to the last quantifiable level (AUC0-t), area under the plasma concentration time curve extrapolated to infinity (AUC0-∞), maximum plasma concentration (Cmax), the plasma elimination half-life (Tmax) and plasma half-life (T1/2) were calculated for both formulations.

DETAILED DESCRIPTION:
Study procedure In each period, the subjects arrived at the clinical/unit site on the day before the commencement of the study and were randomized using Excel® 2007 to receive the test formulation followed by the reference formulation, or viceversa. No food was allowed from 10 h before until at least 4 h after drug administration. On the subsequent morning, a peripheral venous 21G catheter was inserted in the antecubital vein of the subjects and blood samples were collected (zero time). The subjects then received a single 75 mg tablet of either the test or the reference formulation, given with 250 mL water. Blood samples were collected at 0.16, 0.33, 0.5, 0.66, 0.83, 1, 1.5, 1.75, 2, 2.5, 3, 6, 8, 12, 16 and 24 h after drug administration. The blood samples were collected in coded EDTA tubes and plasma was obtained by centrifugation (2,053 g for 10 min at 5 C), after which the plasma was immediately transferred to prelabeled vials and stored at or below -70 After a week of washout, the alternative formulation was administered to the subjects and samples were drawn and analyzed as before.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and age is between 18 and 40 years, inclusive.
2. Females must have negative results for pregnancy tests performed:at Screening on a urine specimen obtained within 2 weeks prior to initial study drug administration, and prior to dosing on urine sample obtained on Study Day -1 of each period
3. Body Mass Index (BMI) is 19 to 26, inclusive. BMI is calculated as weight in kg divided by the square of height measured in meters.
4. A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).
5. Must voluntarily sign and date each informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

1. History of significant sensitivity to any drug.
2. Requirement for any over-the-counter and/or prescription medication, vitamins and/or herbal supplements, on a regular basis.
3. Use of any medications, vitamins and/or herbal supplements, within the 1-week period prior to study drug administration.
4. Pregnant or breastfeeding female.
5. Recent (6-month) history of drug or alcohol abuse.
6. Positive test result for hepatitis B surface antigen (HBsAg) or HIV antibodies (HIV Ab). Negative HIV status will be confirmed at Screening and the results will be maintained confidentially by the study site.
7. Use of known inhibitors (e.g., ketoconazole) or inducers (e.g., carbamazepine) of cytochrome P450 3A (CYP3A) within 1 month prior to study drug administration.
8. Positive screen for drugs of abuse, or alcohol or nicotine or positive and clinically significant urine adulterants test.
9. Receipt of any drug by injection within 30 days or within a period defined by 5 half-lives, whichever is longer, prior to study drug administration.
10. History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
11. History of gastric surgery, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption.
12. Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration.
13. Receipt of any investigational product within 8 weeks prior to study drug administration or 7 half-lives, whichever is longer.
14. Consumption of alcohol within the 3-day period prior to study drug administration.
15. Consumption of grapefruit or grapefruit products, Seville oranges, star fruit and quinine/tonic water from 3 days prior to study drug administration.
16. Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration.
17. Current enrollment in another clinical study.
18. Consideration by the investigator, for an reason, that the subject is an unsuitable candidate to receive Ibuprofen

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration (Cmax) | at 0.16, 0.33, 0.5, 0.66, 0.83, 1, 1.5, 1.75, 2, 2.5, 3, 6, 8, 12, 16 and 24 h after drug administration

SECONDARY OUTCOMES:
area under the plasma concentration time curve from zero to the last quantifiable level (AUC0-t), | 0.16, 0.33, 0.5, 0.66, 0.83, 1, 1.5, 1.75, 2, 2.5, 3, 6, 8, 12, 16 and 24 h after drug administration
area under the plasma concentration time curve extrapolated to infinity (AUC0-∞) | at 0.16, 0.33, 0.5, 0.66, 0.83, 1, 1.5, 1.75, 2, 2.5, 3, 6, 8, 12, 16 and 24 h after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Garza Ocañas, MD PhD, Principal Investigator — Hospital Universitario Jose E Gonzalez
Locations (1):
- Departamento de Farmacologia y Toxicologia, Monterrey, Nuevo León, Mexico